CLINICAL TRIAL: NCT02522429
Title: Thalamic Low Intensity Focused Ultrasound Stimulation in Disorders of Consciousness Following Severe Brain Injury
Brief Title: Thalamic Low Intensity Focused Ultrasound in Brain Injury
Acronym: LIFUP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 restrictions placed on the study.
Sponsor: University of California, Los Angeles (Other)
Collaborators: The Dana Foundation (Other); Tiny Blue Dot Foundation (Other)
Responsible Party: Principal Investigator, Martin M Monti, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 441488-MM-58041
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Consciousness Disorders; Brain Injuries
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries

STUDY DESIGN:
Intervention Model Description: 15 acute DOC patients and 15 chronic DOC patients.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low Intensity Focused Ultrasound Device (Experimental): 15 acute DOC patients, 15 chronic DOC patients
  Interventions: Device: Low Intensity Focused Ultrasound Device

INTERVENTIONS:
Device: Low Intensity Focused Ultrasound Device — Low Intensity Focused Ultrasound Pulsation (LIFUP) of thalamus (a key area for the consciousness network) will be performed during two sessions (one occurring after deep sedation is stopped and the second one occurring just before discharge). The proposed experiment will involve behavioral (i.e., CRS-R) and paramedical (i.e., MRI/fMRI and EEG) measurements just before and after each of the two LIFUP sessions (i.e., 5 non-consecutive minutes of stimulation in each session).
  Other Names: BX Pulsar 1001; BX Pulsar 1002

SUMMARY:
Few neurological conditions are as scientifically mysterious and clinically, legally, and ethically challenging as disorders of consciousness. To date there exists no standard intervention for patients suffering from these devastating conditions. The present project is aimed at evaluating the potential of non-invasive Low Intensity Focused Ultrasound Pulsation (LIFUP) of thalamus (a key area for the consciousness network) as a neurorestorative stimulation for those patients. In this study, LIFUP will be performed during two sessions. The proposed experiment will involve behavioral and paramedical measurements just before and after each of the two LIFUP sessions in a small sample of patients (up to 15 acute and 15 chronic patients) in order to evaluate the feasibility of a full scale clinical trial.

DETAILED DESCRIPTION:
Few neurological conditions are as scientifically mysterious and clinically, legally, and ethically challenging as disorders of consciousness (DOC). Typically developed after severe brain injury, this set of related conditions includes Coma, the Vegetative State (VS) and the Minimally Conscious State (MCS). In the past 20 years, an increasing amount of research has broken many conventions about these disorders, including the once widespread belief that these patients are entirely apallic - that is, lack any kind of "higher" activity. Since then, it has been shown that a lot of brain activity, including relatively high-level cognitive processes, can remain in DOC patients. Nonetheless, to date there exists no standard intervention for patients suffering from these devastating conditions. Developing interventions for this population is extremely important first and foremost for the well-being of patients, who - today - remain completely dependent on assisted care, are often unable to participate in rehabilitative programs because of their lack of behavioral responsiveness, and thus find themselves prisoners of a condition characterized by uncertainty at the medical, legal and ethical decision-making levels. In addition, these conditions, which can last indefinitely, also place great emotional and monetary strain on families, large burdens on care-takers - often leading to increased rates of burn-out - and large financial stress on medical structures and public finances due to the large costs imposed by prolonged intensive care.

The present project is aimed at evaluating the potential of non-invasive Low Intensity Focused Ultrasound Pulsation (LIFUP) of thalamus (a key area for the consciousness network) as a neurorestorative stimulation for patients with severe brain injury.

LIFUP will be performed during two sessions (one occurring after deep sedation is stopped and the second one occurring just before discharge). The proposed experiment will involve behavioral (i.e., CRS-R) and paramedical (i.e., MRI/fMRI) measurements just before and after each of the two LIFUP sessions (i.e., 5 non-consecutive minutes of stimulation in each session) in a small sample of patients (up to 15 acute and 15 chronic DOC patients) in order to evaluate the feasibility of a full scale clinical trial.

The duration of participation in the study will be a year. In terms of impact, we think this project would have a number of immediate consequences. (i) A successful pilot study and any indication that this approach might have the hypothesized effect would place us in a unique position to initiate a fully-fledged double-blind clinical trial in a large cohort of patients.

(ii) From a purely scientific point of view, by virtue of testing what is today the most prominent physiological hypothesis concerning loss and recovery of consciousness after severe brain injury, this project has a direct repercussion on our understanding of the mechanisms underlying these conditions. (iii) From a clinical and patient management point of view the present project is the first necessary step towards opening a completely new avenue for care-taking in patients suffering from this devastating condition for which there is no intervention. In particular, if this project were successful in the long run (e.g., after a double-blind full clinical trial), it could make widely available a non-invasive protocol which could substitute the currently highly invasive (and therefore not widely available, and high risk) only intervention available.

ELIGIBILITY:
Inclusion Criteria:

Acute patients

* < 6 weeks since injury
* a Glasgow Coma Score < 9 (at the time of injury)
* an abnormal CT
* prolonged loss of consciousness (>24h)
* behavioral profile consistent with a VS or MCS as assessed with the Coma Recovery Scale Revised.

Chronic patients:

* > 3 months post injury for non-traumatic injuries, >12 months post-injury for traumatic injuries
* behavioral profile consistent with a VS or MCS as assessed with the Coma Recovery Scale Revised.

Exclusion Criteria (all patients):

* deep sedation
* history of neurological illness prior to injury
* inability to safely enter the MR environment (e.g., ferromagnetic non MR safe implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin M Monti, Prof, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Intensity Focused Ultrasound Device: 15 acute DOC patients, 15 chronic DOC patients
  Low Intensity Focused Ultrasound Device: Low Intensity Focused Ultrasound Pulsation (LIFUP) of thalamus (a key area for the consciousness network) will be performed during two sessions (one occurring after deep sedation is stopped and the second one occurring just before discharge). The proposed experiment will involve behavioral (i.e., CRS-R) and paramedical (i.e., MRI/fMRI) measurements just before and after each of the two LIFUP sessions (i.e., 5 non-consecutive minutes of stimulation in each session).
Period: Overall Study
Arm/Group | Low Intensity Focused Ultrasound Device
Started | 23 (Acute: 13 Chronic: 10)
Completed | 11 (Acute: 4 Chronic: 7)
Not Completed | 12
Not completed — Lost to Follow-up | 8
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Patient exceeded inclusion criteria after enrollment but prior to undergoing study procedures | 1

BASELINE CHARACTERISTICS:
Arm/Group | Low Intensity Focused Ultrasound Device
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] — Population: Reporting separately Acute and Chronic patients
  years
    Acute: number analyzed (Participants) | 13
    Acute | 31 [22 to 75]
    Chronic: number analyzed (Participants) | 10
    Chronic | 35 [26 to 58]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Reporting separately Acute and Chronic patients
  Participants
    Acute: number analyzed (Participants) | 13
    Acute: Female | 2
    Acute: Male | 11
    Chronic: number analyzed (Participants) | 10
    Chronic: Female | 4
    Chronic: Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23
Time Post Injury [Median (Standard Deviation); unit: Days] — Population: Reporting separately Acute and Chronic patients
  Days
    Acute: number analyzed (Participants) | 13
    Acute | 23 (28.32)
    Chronic: number analyzed (Participants) | 10
    Chronic | 1076 (2029)

OUTCOME MEASURES:

1. Primary Outcome: Number of Voxels in Which the Functional Magnetic Resonance Imaging (fMRI) Signal is Significantly Associated to LIFUP Across the Whole Group (Session 1)
Description: Number of voxels found to have a functional MRI signal (measured with a Blood Oxygenation Level Dependent sequence) significantly associated with the onset/offset of the LIFUP stimulation across the tested population.
Time Frame: day 3 (+/-2)
Population: Separating Acute and Chronic patients
Measure: Number; unit: Number of significant voxels
Units Other Than Participants: Voxels
Arm/Group | Low Intensity Focused Ultrasound Device
Number analyzed (Participants) | 21
Number analyzed (Voxels) | 228453
Number of significant voxels
  Acute: number analyzed (Participants) | 11
  Acute | 211
  Chronic: number analyzed (Participants) | 10
  Chronic | 0
Statistical Analysis 1: Comparison: Low Intensity Focused Ultrasound Device; Test type: Other; p = 0.05, t-test, 1 sided — Statistic adjusted at familywise level alpha of 0.05 with a Gaussian Random Field Cluster Correction (Z > 2.7)

2. Primary Outcome: Number of Voxels in Which the Functional Magnetic Resonance Imaging (fMRI) Signal is Significantly Associated to LIFUP (Session 2)
Description: Number of voxels found to have a functional MRI signal (measured with a Blood Oxygenation Level Dependent sequence) significantly associated with the onset/offset of the LIFUP stimulation.
Time Frame: day 10 (+/-2)
Population: Separating Acute and Chronic (including only patients who underwent a second session)
Measure: Number; unit: Number of significant voxels
Units Other Than Participants: Voxels
Arm/Group | Low Intensity Focused Ultrasound Device
Number analyzed (Participants) | 13
Number analyzed (Voxels) | 228453
Number of significant voxels
  Acute: number analyzed (Participants) | 4
  Acute | 0
  Chronic: number analyzed (Participants) | 9
  Chronic | 0
Statistical Analysis 1: Comparison: Low Intensity Focused Ultrasound Device; Test type: Other; p < 0.05, t-test, 1 sided — Statistic adjusted at familywise level alpha of 0.05 with a Gaussian Random Field Cluster Correction (Z > 2.7). All significant voxels have an associated p-value smaller-or-equal to 0.05 (corrected for multiplicity)

3. Primary Outcome: Number of Participants With (Severe) Adverse Events
Description: Number of AEs and SAEs occurring throughout the paradigm.
Time Frame: day 16 (+/-3)
Measure: Number; unit: participants
Arm/Group | Low Intensity Focused Ultrasound Device
Number analyzed (Participants) | 23
participants | 3

4. Secondary Outcome: Coma Recovery Scale Revised (CRS-R)
Description: The Coma Recovery Scale Revised (CRS-R) is a standard clinical protocol specifically developed to assess a patient's level of consciousness, and does so by evaluating a patient's level of responsiveness to sensory stimulation, their ability to understand language, and to communicate. This procedure is typically administered at bedside. The protocol is divided into 6 sub-scales, each assessing a different area (e.g., visual function, auditory function, communication, arousal), and the final score is calculating by adding all sub-scales.The total score of this scale goes from its minimum, 0, which implied a state of coma, to 23, which implies emergence from a Minimally Conscious State (i.e., eMCS). Higher values thus map onto better outcomes.
Time Frame: Change in maximum CRS-R score in the 3 measurements following LIFUP (day of, day after, 1 week after) compared to the maximum CRS-R score in the 3 measurements prior to LIFUP (1 week before, day before, day of).
Population: Reporting separately Acute and Chronic patients; higher scores mean better outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Intensity Focused Ultrasound Device
Number analyzed (Participants) | 21
score on a scale
  Acute: number analyzed (Participants) | 11
  Acute | 2.8 (3.6)
  Chronic: number analyzed (Participants) | 10
  Chronic | 1.5 (2.8)
Statistical Analysis 1: Comparison: Low Intensity Focused Ultrasound Device; Maximum CRS-R prior to LIFUP compared to Maximum CRS-R after LIFUP; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Glasgow Outcome Scale-Extended (GOS-E)
Description: The Glasgow Outcome Scale extended (GOS-E) is a global scale that classifies functional outcome in brain injury patients. Specifically, the scale, which ranges from a minimum total score of 1 (i.e., Dead) to a maximum total score of 8 (Upper Good Recovery), classifies patient status into one of eight categories: Dead (score: 1), Vegetative State (score: 2), Lower Severe Disability (score: 3), Upper Severe Disability (score: 4), Lower Moderate Disability (score: 5), Upper Moderate Disability (score: 6), Lower Good Recovery (score: 7), or Upper Good Recovery (score: 8). Higher scores thus represent better outcomes. The score is determined according to specific answers given in the instrument.
Time Frame: day 16 (+/-3) and day 180 (+/-15)
Population: Separating Acute (7/11 lost to 14 day follow up; 9/11 lost to 6-month follow-up [including COVID19 restrictions]) and Chronic groups (1/10 lost to 14 day follow-up; 3/10 lost to 6-month follow-up [including COVID19 restrictions])
Measure: Median (Full Range); unit: score on a scale (higher scores better)
Arm/Group | Low Intensity Focused Ultrasound Device
Number analyzed (Participants) | 13
score on a scale (higher scores better)
  Acute (14-day follow-up): number analyzed (Participants) | 4
  Acute (14-day follow-up) | 3 [2 to 3]
  Chronic (14-day follow-up): number analyzed (Participants) | 9
  Chronic (14-day follow-up) | 3 [2 to 3]
  Acute (6-month follow-up): number analyzed (Participants) | 2
  Acute (6-month follow-up) | 3 [3 to 3]
  Chronic (6-month follow-up): number analyzed (Participants) | 7
  Chronic (6-month follow-up) | 3 [2 to 3]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Low Intensity Focused Ultrasound Device
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Intensity Focused Ultrasound Device (N=23)
Respiratory depression (prior to any intervention procedure) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Early termination due to COVID-19 imposed restrictions prevented acquisition of intended sample and follow-up data for a majority of patients.
2. Length of the protocol on each exposure session prevented acquisition of the originally planned structural MRI (for Primary outcomes #1, #3) and the EEG data before/after exposure (for Secondary outcome #2).
3. Loss of majority of Acute patients to follow-up prevents meaningful group analysis for Primary outcome #4 in the Acute cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT02522429/Prot_SAP_000.pdf